CLINICAL TRIAL: NCT03599830
Title: Study of the Cognition of Patients Treated With
Brief Title: Study of the Cognition of Patients Treated With Immunotherapy
Acronym: COG-IMMUNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A01041-54
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Patients With Cancer Who Start Immunotherapy; All Neoplasms
Keywords: Immunotherapy; Cognition; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive test passations (Other): 3 neuropsychological passations over a period of 6 months.
  Interventions: Other: Cognitive test passations

INTERVENTIONS:
Other: Cognitive test passations — Tests :
  MoCA2 Hopkins verbal learning test WAIS-IV Trail Making test Stroop Verbal fluences

SUMMARY:
The investigator's longitudinal pilot study aims to evaluate for the first time the impact of immunotherapy on cognition in oncology.

Due to the recent nature of immunotherapy, its side effects and impact on quality of life are still poorly understood and, to date, there is no published study evaluating the impact of immunotherapy on cognition in patients treated for cancer.

The study consists of the passation of 3 neuropsychological assessments over a period of 6 months in cancer patients who start immunotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18,
* Patient with cancer and having to initiate treatment with immunotherapy alone
* Treatment with immunotherapy will include either an anti-PD1 / L1 or Anti CTLA4 monotherapy or combination,
* Patients may have received other antitumor treatments other than immunotherapy but these should be stopped at the time of initiation of immunotherapy
* Performance Status <2
* Patient at the level of studies 3 "end of primary studies" minimum (Barbizet scale),
* Mastery of the French language.
* Patient affiliated to a social security system
* Patient having attested in writing of his non-opposition to participate in the study

Exclusion Criteria:

* Previous treatment with immunotherapy
* Another anti-tumor treatment underway
* Primary cancer of the central nervous system or cerebral metastasis, symptomatics and not controlled
* Abuse of alcohol or drug use
* Severe visual and / or auditory deficiency,
* Refusal of participation of the patient.
* Patient deprived of liberty or under guardianship
* Patient unable to follow the study for geographical, social or psychopathological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function (at least in a cognitive domain) | between inclusion and 3 months.
  The proportion of patients who will have a reduction of scores in neuropsychological questionnaires (scores of MoCA2, Hopkins verbal learning test, WAIS-IV, Trail Making test, Stroop Symboles)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Chu Amiens, Amiens
  - CHU CAEN, Caen
  - Centre François Baclesse, Caen
  - Chru Lille, Lille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lange M, Clarisse B, Leconte A, Dembele KP, Lequesne J, Nicola C, Dubois M, Derues L, Gidron Y, Castel H, Joly F. Cognitive assessment in patients treated by immunotherapy: the prospective Cog-Immuno trial. BMC Cancer. 2022 Dec 13;22(1):1308. doi: 10.1186/s12885-022-10384-y. PMID 36513991